CLINICAL TRIAL: NCT04809454
Title: Frequency of Florid Hyperthyroidism In Patients Taking Iodinated Salt: A Cross Sectional Study
Brief Title: Frequency of Florid Hyperthyroidism In Patients Taking Iodinated Salt
Acronym: I2 and thyroid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Mehwish Iftikhar, Principal Investigator, Services Institute of Medical Sciences, Pakistan
Other Study IDs: 1241985
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Thyroid Dysfunction
Keywords: Thyroid; Iodine
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroxin a vital hormone for life lot of body functions depend on proper functioning on pituitary thyroid axis. it exists in two major forms Thyroxine (T4) and (T3) , each of them containing two iodine atoms on their inner (tyrosine) ring. Synthesis of reasonable quantities of thyroid hormones requires adequate iodine intake to allow sufficient thyroidal uptake. The World Health Organization (WHO) recommendation for daily intake of iodine is 150 μg for children ≥12 years and adults, and 250 μg for pregnant and lactating women. However as we know optimum amount of iodine is required for normal pituitary thyroid axis like wise excessive intake may cause over functioning of axis hence over production of hormone that can be manifested both clinically and biochemically.

This study is designed to observe the frequency of over hyperthyroidism in patients taking iodinated salt.

DETAILED DESCRIPTION:
All patients presenting to endocrine clinic fulfilling inclusion and exclusion criteria will be recruited. They will be examined, their vitals including blood pressure pulse will be noted, thyroid clinical examination including eye signs and thyroid status will be done biochemical Thyroid profile (TSH, Free T3 & Free T4) will be noted in predesigned proforma.

Statistical Analysis will be done ,after data is entered in Statistical Package for the Social Sciences (SPSS) version 25 .qualitative data will be presented as frequencies and percentages while quantitative data will be presented as mean medians and standard deviations.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presenting with biochemical hyperthyroidism
2. Who are taking Iodinated salt.
3. Treatment naïve patients
4. Both genders included
5. All patients who can give consent (18-60 years)

Exclusion Criteria:

1) Pregnant females 2) Lactating mothers

-

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All patients presenting with biochemical hyperthythyroidism and taking Iodinated salt with age range of 18-60 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Affect of Iodinated Salt on Thyroid Status | through study completion an average of 12 weeks
  Affect of Iodinated Salt on Thyroid Status

CONTACTS AND LOCATIONS:
Locations (1):
- Mehwish Iftikhar, Lahore, Punjab Province, Pakistan